CLINICAL TRIAL: NCT05374278
Title: First-in-Human Evaluation of an Astrocytic Glutamate Transporter (EAAT2) PET Tracer in the Brains of Healthy Controls and Patients With Dementia.
Brief Title: First-in-Human Evaluation of an Astrocytic Glutamate Transporter (EAAT2) PET Tracer in Dementia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David Wilson (Other)
Collaborators: Rio pharmaceuticals Inc. (Unknown)
Responsible Party: Sponsor-Investigator, David Wilson, Professor, Radiology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13180640
Record Dates: First submitted 2021-12-24; First posted 2022-05-16 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Frontotemporal Dementia; Dementia
Keywords: Alzheimer Disease; Nuclear medicine; Positron emission tomography; Magnetic resonance imaging; Frontotemporal Dementia
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia; Dementia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 - dosimetry of [18F]RP-115 in healthy volunteers (Experimental): Establish [18F]RP-115 safety in the clinic with male and female PET imaging.
  Interventions: Drug: [18F]RP-115 PET/MRI or PET/CT and MRI
- Cohort 2B - [18F]RP-115 in patients with AD (Experimental): Comparison of [18F]RP-115 PET binding between AD patients and age-matched cognitively normal controls and between AD and FTD
  Interventions: Drug: [18F]RP-115 PET/MRI or PET/CT and MRI
- Cohort 2C - [18F]RP-115 in patients with FTD (Experimental): Comparison of [18F]RP-115 PET binding between AD patients and age-matched cognitively normal controls and between AD and FTD
  Interventions: Drug: [18F]RP-115 PET/MRI or PET/CT and MRI
- Cohort 2A - [18F]RP-115 in age-matched controls (Experimental): Comparison of [18F]RP-115 PET binding between AD patients and age-matched cognitively normal controls and between AD and FTD
  Interventions: Drug: [18F]RP-115 PET/MRI or PET/CT and MRI

INTERVENTIONS:
Drug: [18F]RP-115 PET/MRI or PET/CT and MRI — An I.V. bolus injection of up to 10 millicurie (mCi) [18F]RP-115 will be administered, followed by a PET/MRI scan or by a combination of PET/CT and MRI

SUMMARY:
This is a first in human study that will assess the safety and diagnostic performance of [18F]RP-115 (fluorine-18 labeled RP115), a positron emission tomography (PET) agent. This agent has the potential to identify the early changes that occur in the brains of patients with Alzheimer's disease (AD) and frontotemporal dementia (FTD).

DETAILED DESCRIPTION:
AD and FTD are the two leading causes of dementia with tremendous impact on patients and their families. Early diagnosis of both AD and FTD is essential to increase patients' quality of life, identify and treat reversible causes, and enhance the development and effectiveness of treatments. However, no single diagnostic agent is currently available for either AD or FTD; instead, clinicians must rely on the patient's history and cognitive testing which often leads to delayed or incorrect diagnosis. Importantly AD and FTD have distinct regional patterns of neuronal loss and dysfunction in the brain; an agent that could detect these regionally specific changes early in the course of the disease process could revolutionize diagnosis and treatment development for these conditions.

This study aims to develop a novel radiotracer to fill this unmet need. The excitatory amino acid transporter 2 (EAAT2) is the main transporter for glutamate in the brain and has been shown to be downregulated in the context of AD and other neurodegenerative conditions. EAAT2 is responsible for over 90% of glutamate uptake in the brain where it is primarily located on astrocytes and plays a key role in maintaining the homeostasis of the tripartite synapse. The goal of this study is to test the EAAT2 targeted positron emitting agent, [18F]RP-115, to evaluate early changes in astrocytes in healthy controls versus patients with AD and FTD by quantitative PET imaging of EAAT2. We have preclinical data that demonstrates that this agent is a good predictor of EAAT2 levels in animal models, hence, can potentially detect early signs of neurodegeneration. We now wish to test this agent in humans.

In summary, the primary objective of this study is to demonstrate human safety and measure the biodistribution of [18F]RP-115 in healthy controls as well as in age-matched patients with AD and FTD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-75
2. Age-suitable BMI
3. Ability to provide written informed consent and willingly comply with protocol requirements or has a legal authorized representative/guardian who provides surrogate informed consent.
4. No apparent physical disorder.
5. Radial, ulnar, or brachial artery suitable for catheterization.
6. Non-smoker, and not taking OTC nicotine cessation - to limit peripheral metabolism events.
7. Devoid of CNS prescription drugs for three weeks - to limit peripheral metabolism events.

   For Cohort 2B and 2C:
8. Must have a study partner (informant) who spends a minimum average of 5 hours per week with the participant (e.g. family member, significant other, friend, caregiver), is generally aware of the participant's daily activities, can provide information about the participant's cognitive and functional performance, and will accompany the participant in all study procedure.
9. Recent (within 6 mo.) MME clinical scores.

Exclusion Criteria:

1. Unable to provide written informed consent and unwilling to comply with protocol requirements, or does not have a legal authorized representative/guardian who can provide surrogate informed consent.
2. Inadequate arterial access.
3. Receipt of radioisotope < 5 half-lives within [18F]RP-115 imaging- as to not confound any scans with radiation background for previous scanning, and unsuitable organ dosimetry thresholds from previous (> two weeks) PET scans.
4. The performed [18F]RP-115 scan(s) must not represent > 3 PET studies total within one year.
5. Contra-indication to magnetic resonance, including permanent pacemaker, implantable metallic device, etc.; or severe claustrophobia.
6. Participants who are pregnant (female patients of childbearing age will be tested prior to injection of tracer- positive test excludes from the study)
7. Participants who are breast-feeding.
8. Have a medical condition or other circumstances that in the opinion of the project physicians would significantly decrease chances of obtaining reliable data, achieving the study objective or completing the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2027-04-03 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety of Administered dose | A year
  Each study participant will undergo a physical examination, vital signs, and ECGs prior to and after the scan and will also be monitored during the scan for adverse events. Additionally, a follow-up with the subject will be conducted 24-48 hours after [18F]RP-115 administration.
  Outcome Measure: Any adverse events will be recorded and graded according to Common Terminology Criteria for Adverse Events.
Dosimetry of [18F]RP-115 | A year
  Whole-body PET/MRI scan will be conducted immediately after an [18F]RP-115 injection and last about 3.5 hours (including breaks) in 8 healthy volunteers (male and female). Equivalent organ radiation doses will be calculated in selected organs using the dynamic PET/MRI data in order to calculate the dosimetry of the tracer.
  Outcome Measure: Radiation exposure per organ as milliSievert/kg
Biodistribution of [18F]RP-115 | A year
  Whole-body PET/MRI scan will be conducted immediately after an [18F]RP-115 injection and last about 3.5 hours (including breaks) in 8 healthy volunteers (male and female). Percent injected activity (%IA) will be calculated in selected organs using the dynamic PET/MRI data in order to calculate the biodistribution of the tracer.
  Outcome Measure: Percent injected activity (%Injected radioactivity) in selected organs.

SECONDARY OUTCOMES:
[18F]RP-115 diagnostic performance | Three years
  Utilize RP-115 to quantitatively assess regional cerebral RP-115 binding differences in healthy volunteers compared to cognitively-defined AD and FTD.
  Outcome Measure: Radioactivity distribution volume across cerebral cortex, Becquerel/mL or standardized uptake value.

CONTACTS AND LOCATIONS:
Overall Officials: David Wilson, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- China Basin, UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individuals participants data collected during the trial, after de-identification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data

REFERENCES:
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606
- [Background] Boche D, Gerhard A, Rodriguez-Vieitez E; MINC Faculty. Prospects and challenges of imaging neuroinflammation beyond TSPO in Alzheimer's disease. Eur J Nucl Med Mol Imaging. 2019 Dec;46(13):2831-2847. doi: 10.1007/s00259-019-04462-w. Epub 2019 Aug 8. PMID 31396666
- [Background] Innis RB, Cunningham VJ, Delforge J, Fujita M, Gjedde A, Gunn RN, Holden J, Houle S, Huang SC, Ichise M, Iida H, Ito H, Kimura Y, Koeppe RA, Knudsen GM, Knuuti J, Lammertsma AA, Laruelle M, Logan J, Maguire RP, Mintun MA, Morris ED, Parsey R, Price JC, Slifstein M, Sossi V, Suhara T, Votaw JR, Wong DF, Carson RE. Consensus nomenclature for in vivo imaging of reversibly binding radioligands. J Cereb Blood Flow Metab. 2007 Sep;27(9):1533-9. doi: 10.1038/sj.jcbfm.9600493. Epub 2007 May 9. PMID 17519979
- [Background] Rice L, Bisdas S. The diagnostic value of FDG and amyloid PET in Alzheimer's disease-A systematic review. Eur J Radiol. 2017 Sep;94:16-24. doi: 10.1016/j.ejrad.2017.07.014. Epub 2017 Jul 20. PMID 28941755
- [Background] Rodriguez-Vieitez E, Carter SF, Chiotis K, Saint-Aubert L, Leuzy A, Scholl M, Almkvist O, Wall A, Langstrom B, Nordberg A. Comparison of Early-Phase 11C-Deuterium-l-Deprenyl and 11C-Pittsburgh Compound B PET for Assessing Brain Perfusion in Alzheimer Disease. J Nucl Med. 2016 Jul;57(7):1071-7. doi: 10.2967/jnumed.115.168732. Epub 2016 Feb 16. PMID 26912447
- [Background] Arakawa R, Stenkrona P, Takano A, Nag S, Maior RS, Halldin C. Test-retest reproducibility of [11C]-L-deprenyl-D2 binding to MAO-B in the human brain. EJNMMI Res. 2017 Dec;7(1):54. doi: 10.1186/s13550-017-0301-4. Epub 2017 Jun 20. PMID 28634836
- [Background] Cowburn R, Hardy J, Roberts P, Briggs R. Presynaptic and postsynaptic glutamatergic function in Alzheimer's disease. Neurosci Lett. 1988 Mar 21;86(1):109-13. doi: 10.1016/0304-3940(88)90192-9. PMID 2896322
- [Background] Scott HL, Tannenberg AE, Dodd PR. Variant forms of neuronal glutamate transporter sites in Alzheimer's disease cerebral cortex. J Neurochem. 1995 May;64(5):2193-202. doi: 10.1046/j.1471-4159.1995.64052193.x. PMID 7722505
- [Background] Hoshi A, Tsunoda A, Yamamoto T, Tada M, Kakita A, Ugawa Y. Altered expression of glutamate transporter-1 and water channel protein aquaporin-4 in human temporal cortex with Alzheimer's disease. Neuropathol Appl Neurobiol. 2018 Oct;44(6):628-638. doi: 10.1111/nan.12475. Epub 2018 Mar 4. PMID 29405337
- [Background] Li S, Mallory M, Alford M, Tanaka S, Masliah E. Glutamate transporter alterations in Alzheimer disease are possibly associated with abnormal APP expression. J Neuropathol Exp Neurol. 1997 Aug;56(8):901-11. doi: 10.1097/00005072-199708000-00008. PMID 9258260
- [Background] Pasqualetti G, Brooks DJ, Edison P. The role of neuroinflammation in dementias. Curr Neurol Neurosci Rep. 2015 Apr;15(4):17. doi: 10.1007/s11910-015-0531-7. PMID 25716012
- [Background] Miller ZA, Sturm VE, Camsari GB, Karydas A, Yokoyama JS, Grinberg LT, Boxer AL, Rosen HJ, Rankin KP, Gorno-Tempini ML, Coppola G, Geschwind DH, Rademakers R, Seeley WW, Graff-Radford NR, Miller BL. Increased prevalence of autoimmune disease within C9 and FTD/MND cohorts: Completing the picture. Neurol Neuroimmunol Neuroinflamm. 2016 Oct 28;3(6):e301. doi: 10.1212/NXI.0000000000000301. eCollection 2016 Dec. PMID 27844039
- [Background] Arnold SE, Han LY, Clark CM, Grossman M, Trojanowski JQ. Quantitative neurohistological features of frontotemporal degeneration. Neurobiol Aging. 2000 Nov-Dec;21(6):913-9. doi: 10.1016/s0197-4580(00)00173-1. PMID 11124442
- [Background] Lui H, Zhang J, Makinson SR, Cahill MK, Kelley KW, Huang HY, Shang Y, Oldham MC, Martens LH, Gao F, Coppola G, Sloan SA, Hsieh CL, Kim CC, Bigio EH, Weintraub S, Mesulam MM, Rademakers R, Mackenzie IR, Seeley WW, Karydas A, Miller BL, Borroni B, Ghidoni R, Farese RV Jr, Paz JT, Barres BA, Huang EJ. Progranulin Deficiency Promotes Circuit-Specific Synaptic Pruning by Microglia via Complement Activation. Cell. 2016 May 5;165(4):921-35. doi: 10.1016/j.cell.2016.04.001. Epub 2016 Apr 21. PMID 27114033
- [Background] Yin F, Banerjee R, Thomas B, Zhou P, Qian L, Jia T, Ma X, Ma Y, Iadecola C, Beal MF, Nathan C, Ding A. Exaggerated inflammation, impaired host defense, and neuropathology in progranulin-deficient mice. J Exp Med. 2010 Jan 18;207(1):117-28. doi: 10.1084/jem.20091568. Epub 2009 Dec 21. PMID 20026663

DOCUMENTS (1):
  • Informed Consent Form (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT05374278/ICF_000.pdf